CLINICAL TRIAL: NCT06338111
Title: Can we Improve Mortality Prediction in Patients With Sepsis in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Sonia Luka, Teaching Assistant PhD Student Sonia Luka, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 2461
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Sepsis Syndrome; Emergency Department; Biomarker
Keywords: Procalcitonin; Azurocidin 1; High Sensitivity C reactive protein; Urokinase-type plasminogen activator system; Soluble triggering receptor expressed on myeloid cells - 1; Interleukin-6; Severity scores; Emergency Department; Sepsis; Septic shock
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Emergencies; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biochemistry blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 09.11.2020-01.08.2021, patients with sepsis and septic shock
  Interventions: Diagnostic Test: ELISA Sepsis Biomarkers dosage
- 2: 13.07.2022-04.12.2022, patients with sepsis and septic shock
  Interventions: Diagnostic Test: ELISA Sepsis Biomarkers dosage

INTERVENTIONS:
Diagnostic Test: ELISA Sepsis Biomarkers dosage — Observational
  Other Names: ELISA Specific Sepsis Biomarkers dosage

SUMMARY:
This study aims to identify the prognostic role of procalcitonin (PCT), soluble Triggering Receptor Expressed on Myeloid Cells-1 (sTREM-1), the soluble form of the urokinase plasminogen activator receptor (suPAR), highly sensitive C-reactive protein (hs-CRP), Interleukin-6 (IL-6), and azurocidin 1 (AZU1) in 28-day mortality for patients with sepsis in Emergency Department.

DETAILED DESCRIPTION:
The levels of the specified biomarkers were measured upon patient arrival at the Emergency Department (ED) and analyzed their correlation with 28-day mortality. The values of these biomarkers were monitored over the initial three days following admission to the ED, aiming to explore their potential in guiding the de-escalation of antibiotic treatment. Considering their prognostic significance, the main goal is to develop a novel scoring system tailored for use in the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis 3 Criteria

Exclusion Criteria:

* individuals aged under 18 or above 90
* pregnant women
* individuals in custody or deprived of their liberty
* patients with associated pathologies such as severe trauma
* other types of shocks
* acute stroke
* burns
* pancreatitis myocardial infarction, pulmonary edema, status asthmatics, convulsions, drug overdose, those requiring emergency surgery
* terminal stage of neoplastic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis or septic shock patients admitted to ED
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Can we better predict mortality in septic patients from the Emergency Department? | 03.2024-05.2024
  Evaluation of the prognostic role of : IL-6, sTREM-1, suPAR, AZU1, hsPCR and PCT in predicting 28-day mortality in Emergency Department

CONTACTS AND LOCATIONS:
Locations (1):
- Cluj County Hospital Emergency Department, Cluj-Napoca, Cluj, Romania